CLINICAL TRIAL: NCT02437812
Title: A Phase II, Open-Label, Non-Randomized, Pilot Study of Paclitaxel, Carboplatin and Oral Metformin for Patients Newly Diagnosed With Stage II-IV Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Study of Paclitaxel, Carboplatin and Oral Metformin in the Treatment of Advanced Stage Ovarian Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gynecologic Oncology Associates (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOA-TCOM1
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-08

CONDITIONS: Epithelial Ovarian Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Metformin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, carboplatin and metformin (Experimental): Drug: Metformin (850 mg) Drug: Carboplatin (AUC 5 or 6) Drug: Paclitaxel (80 mg/m2)
  The regimen will be administered as a dose dense schedule.
  Interventions: Drug: Metformin; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Metformin — Metformin with standard chemotherapy
  Other Names: Glucophage
Drug: Paclitaxel — Standard chemotherapy
  Other Names: Taxol
Drug: Carboplatin — Standard chemotherapy
  Other Names: Carbo

SUMMARY:
Initially, the prospect of metformin as a neoplastic treatment was considered for malignancies of the prostate, colon and pancreas. However, only select clinical studies involving the use of metformin in the treatment of ovarian cancer have documented improved survival rates. Since no first line regimen has demonstrated compelling superiority in the management of advanced stage ovarian carcinoma, the combination of paclitaxel, carboplatin, and metformin is of particular interest given the triplet's prospect for achieving increased synergy without compromising patient tolerability.

DETAILED DESCRIPTION:
A phase II, open-label, non-randomized, pilot study assessing the safety, toxicity, and progression free survival of advanced stage ovarian carcinoma patients who underwent treatment with paclitaxel, carboplatin and metformin. An estimated 30 patients will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

Female Gender

Age greater than 18 years

Advanced stage epithelial ovarian, fallopian tube, or primary peritoneal cancer

Adequate bone marrow function

ECOG performance score of 2 or greater

Patients must be able to swallow oral medication.

Exclusion Criteria:

Subjects must NOT be taking metformin or have been on metformin in the past 6 months.

Subjects with a diagnosis of epithelial ovarian, fallopian tube or peritoneal cancers of low malignant potential (borderline carcinomas)

Subjects with concomitant malignancy or a previous malignancy within the past three years, melanoma skin cancer excepted

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-10 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  The primary outcome of progression free survival will compare the percentage of those who have either progressed or died at 1 year with those who were at risk for at least 1 year.

SECONDARY OUTCOMES:
Metabolic biomarker evaluation | 3 months
  Glucose (mg/dL)
Metabolic biomarker evaluation | 3 months
  Fasting insulin (mIU/L)
Metabolic biomarker evaluation | 3 months
  BMI (kg/m2)
Metabolic biomarker evaluation | 3 months
  Urine (mOsm/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa N Abaid, M.D., M.P.H., Principal Investigator — Gynecologic Oncology Associates
Locations (1):
- Gynecologic Oncology Associates, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once all data is reviewed